CLINICAL TRIAL: NCT05044806
Title: Effect of Perioperative Ultrasound-guided Remote Ischemic Conditioning on Myocardial Injury in Acute Myocardial Infarction Patients Undergoing Percutaneous Coronary Intervention: a Prospective Cohort Study
Brief Title: Effect of Perioperative Ultrasound-guided Remote Ischemic Conditioning on Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yu Zheng, Attending doctor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIC
Record Dates: First submitted 2021-09-01; First posted 2021-09-16 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Remote ischemic conditioning; Percutaneous coronary intervention; Infarction; Myocardial injury; Acute myocardial infarction
MeSH Terms: conditions — Infarction | interventions — Percutaneous Coronary Intervention; Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasound-guided-RIC group (Experimental): Patients in the ultrasound-guided-RIC group will receive percutaneous coronary intervention (PCI), usual pharmacotherapy and pre-, per-, and post-operative ultrasound-guided remote ischemic conditioning (RIC). The pressure applied during cuff inflation is total occlusion pressure (TOP) determined with ultrasound measurement.
  Interventions: Other: Ultrasound-guided remote ischemic conditioning; Procedure: Percutaneous coronary intervention
- Traditional RIC group (Experimental): Patients in the traditional RIC group will receive PCI, usual pharmacotherapy and pre-, per-, and post-operative traditional RIC. The pressure applied during cuff inflation is 20 mmHg above systolic blood pressure.
  Interventions: Other: Traditional remote ischemic conditioning; Procedure: Percutaneous coronary intervention
- Control group (Other): Patients in the control group will receive PCI and usual pharmacotherapy.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Other: Ultrasound-guided remote ischemic conditioning — Before conducting RIC, Doppler ultrasound was used to measure the total occlusion pressure (TOP) of brachial artery, which was then determined as the cuff inflation pressure during RIC. The RIC program encompasses four main components of (1) three cycles of remote ischemic pre-conditioning which will be delivered right after the eligibility check and informed consent form signature before PCI; (2) one cycle of remote ischemic per-conditioning, which will be delivered during PCI; (3) three cycles of remote ischemic post-conditioning, which will be delivered within 10 min after PCI; and (4) two sessions per day of remote ischemic post-conditioning which will start on post-operative day 1 and last till hospital discharge. The remote ischemic pre- and post-conditioning share the RIC protocol, which comprises three 3 min cycles of RIC with 3 min intervals of reperfusion in between, while only one single 3 min cycle will be delivered for the remote ischemic per-conditioning.
  Arms: Ultrasound-guided-RIC group
Other: Traditional remote ischemic conditioning — The RIC program encompasses four main components of (1)three cycles of remote ischemic pre-conditioning which will be delivered right after the eligibility check and informed consent form signature before PCI; (2)one cycle of remote ischemic per-conditioning, which will be delivered during PCI; (3)three cycles of remote ischemic post-conditioning, which will be delivered within 10 min after PCI; and (4) two sessions per day of remote ischemic post-conditioning which will start on post-operative day 1 and last till hospital discharge. The remote ischemic pre- and post-conditioning share the RIC protocol, which comprises three 3 min cycles of upper limb ischemia on the arm that is opposite to the PCI side with 3 min intervals of reperfusion in between delivered by an automated cuff inflation/deflation device, while only one single 3 min cycle will be delivered for the remote ischemic per-conditioning. The pressure applied during cuff inflation is 20 mmHg above systolic blood pressure.
  Arms: Traditional RIC group
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention (PCI) will be performed by a cardiologist or doctor who specializes in the heart to open coronary arteries that are narrowed or blocked by the buildup of atherosclerotic plaque. PCI requires cardiac catheterization, which is the insertion of a catheter tube, and live x rays helping to guide the catheter into the heart to inject special contrast dye that will highlight the blockage. To open a blocked artery, another catheter will be inserted over a guidewire, a balloon will be inflated at the tip of that catheter, and a small mesh tube called a stent may be put in the artery to help keep the artery open. After PCI, the catheters will be removed, the opening on the wrist or groin will be closed and bandaged.
  Other Names: coronary angioplasty

SUMMARY:
Acute myocardial infarction (AMI) is an event of myocardial necrosis caused by myocardial ischemia. Although the incidence and economic burden of AMI has declined in high-income countries, the incidence rate of AMI in China has increased dramatically over the past several decades. Initial medical therapy combined with primary percutaneous coronary intervention (PCI) is currently the most important advance in restoring coronary perfusion. Timely reperfusion therapy may halt the progress of necrosis and preserve viable tissue; however, it can also induce myocardial injury and cause cardiomyocyte death, a phenomenon called myocardial ischemia reperfusion injury (IRI), which can increase final myocardial infarct size by up to 50%. Unfortunately, there is no effective intervention for preventing IRI to date, though an improved understanding of the pathophysiology of IRI has led to the suggestion of several innovative therapeutic strategies with the potential for reducing unintended negative side effects of reperfusion therapy in AMI patients. Whether there is a therapeutic intervention that can effectively and safely reduce myocardial infarct size and cardiac mortality has been intensely explored over the years. Against this backdrop, a phenomenon called remote ischemic conditioning (RIC) has long been discussed as a potential approach to address the above issues. The purpose of present study is to investigate the efficacy of perioperative remote ischemic conditioning delivered at individual timepoints (e.g., pre-, per- and post-PCI) on myocardial injury in patients with AMI.

DETAILED DESCRIPTION:
RIC refers to a cardio-protective effect induced by non-invasively applying cycles of physiological ischemia and reperfusion to remote body parts, e.g., through application of a blood pressure cuff or similar device to a remote limb. The actual molecular biological mechanisms underlying RIC may be attributed to a neuro-hormonal pathway conveying a cardio-protective signal from a local limb to the remote heart. The safety of RIC delivered at a single time point (e.g., pre-, per- or post-PCI) in AMI patients has been well established in a number of clinical trials. However, the RIC's cardio-protective effects remain under debate, especially for RIC programs delivered at individual timepoints during operative period (pre-, per- and post-PCI). Besides, in these trials, the cuff compression pressure of RIC protocol is mostly 200mmHg or 20-50mmHg above systolic pressure. Peripheral vascular ischemia effects of upper limbs are different under different pressure conditions. However, no study has been conducted to investigate the clinical effects of RIC training under different pressure conditions. In the present study, ultrasound is used to determine the brachial artery total occlusion pressure (TOP), which is regarded as optimal pressure of flow restriction in ischemic exercise training. And patients in the ultrasound-guided RIC group will receive RIC applying TOP as cuff compression pressure, while compression pressure applied in traditional RIC group patients is 20mmHg above systolic pressure. The purpose of present study is to investigate the effect of perioperative RIC delivered across the full disease cycle, and compare the effects of ultrasound-guided RIC protocol and traditional RIC protocol on cardiac enzyme infarct size, cardiac function, cardiopulmonary endurance and quality of life in patients with AMI.

ELIGIBILITY:
Inclusion Criteria:

1. Newly developed ST segment elevation myocardial infarction (STEMI) and non-ST segment elevation myocardial infarction (non-STEMI) according to clinical symptoms, ECG and laboratory confirmation;
2. Patients aged 18-80 yr;
3. Scheduled for PCI;
4. With normal cognitive function indicated by MMSE score >16 and able to cooperate with intervention;
5. Agreed to participate and signed the consent form.

Exclusion Criteria:

1. Previous STEMI or non-STEMI;
2. Previous coronary artery bypass grafting (CABG) ;
3. Developed thrombolysis within the last 30 days;
4. Cardiogenic shock history;
5. Persistent atrial fibrillation history;
6. Severe complications (e.g. ventricular septal rupture, free wall rupture or acute severe mitral regurgitation) warrant surgical interventions;
7. Uncontrolled hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg);
8. With peripheral neuropathy, peripheral artery disease, superficial thrombophlebitis or deep vein thrombosis;
9. Other severe systemic diseases;
10. Participated in other trials previously.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Infarct size | During 0-72 hours after surgery
  Cardiac enzyme infarct size is assessed as 72-hour area under the curve (AUC) cardiac troponin T (cTnT) release.

SECONDARY OUTCOMES:
Plasma concentration of myocardial infarction-related key biomarkers (PCMIKB) | Three days after surgery
  PCMIKB will be reflected with concentration of cardiac troponin T (cTnT).
B-type natriuretic peptide （BNP） | Three days after surgery
  The concentration of BNP will be measured during perioperative period.
Left ventricular ejection fraction (LVEF) | One week after surgery
  Left ventricular ejection fraction (LVEF) will be measured with two dimensional echocardiography.
Left ventricular end-diastolic volume (LVEDV) | One week after surgery
  Left ventricular end-diastolic volume (LVEDV) will be measured with two dimensional echocardiography.
Left ventricular end systolic volume (LVESV). | One week after surgery
  Left ventricular end systolic volume (LVESV) will be measured with two dimensional echocardiography.
Cardiopulmonary endurance | Three days after surgery
  Cardiopulmonary endurance will be measured with the 6-min walking test (6MWT).
Blood pressure | When postoperative RIC is finished（within 10 minutes after PCI）
  Systolic and diastolic blood pressure will be monitored before and after training.
Heart rate | When postoperative RIC is finished（within 10 minutes after PCI）
  Heart rate will be monitored before and after training.
Total hospital length of stay (LOS) | Up to 1 month
  LOS accounts for total hospital LOS in both acute hospital and rehabilitation hospital after PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Lu, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China